CLINICAL TRIAL: NCT03431974
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Trial to Establish the Efficacy and Safety of Once-Weekly Oral Aminopterin for the Treatment of Subjects With Moderate-To-Severe Psoriasis
Brief Title: Once-Weekly Oral Aminopterin for the Treatment of Subjects With Moderate-To-Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syntrix Biosystems, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMT-PSO-201; 5U44AI114473 (NIH)
Record Dates: First submitted 2018-02-01; First posted 2018-02-13 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Psoriasis
Keywords: Anti-folate
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Over-encapsulated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LD-Aminopterin oral capsule (Experimental): LD-Aminopterin tablets (0.5 mg tablet) over-encapsulated, 3.0 mg (6 tablets) once orally each week for 14 weeks (14 doses).
  Interventions: Drug: LD-Aminopterin oral capsule
- Placebo oral capsule (Placebo Comparator): Placebo capsules containing microcrystalline once orally each week for 14 weeks (14 doses).
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: LD-Aminopterin oral capsule — anti-folate treatment
  Other Names: racemic 4-Aminopteroylglutamic acid; racemic 4-Aminofolic acid
  Arms: LD-Aminopterin oral capsule
Drug: Placebo oral capsule — Microcrystalline filled capsule to mimic capsule containing aminopterin tablets
  Other Names: Placebo (for aminopterin)
  Arms: Placebo oral capsule

SUMMARY:
This study evaluates the treatment of psoriasis with aminopterin. Participants will be treated for 14 weeks with either aminopterin or placebo followed. The participants will not know if they are being treated with aminopterin or placebo.

DETAILED DESCRIPTION:
A Phase 2, multi-center, randomized, double-blind, placebo-controlled study enrolling subjects with moderate-to-severe psoriasis to investigate the safety and efficacy of LD-aminopterin (AMT) (3 mg (six 0.5 mg tablets). Forty-six subjects will be randomized to one of two parallel treatment arms: LD-AMT (3 mg) or placebo, in a 1:1 ratio. The endpoint analysis will include efficacy and safety. Randomized subjects will initially enter a 14-week treatment phase, followed by a 6-week post-treatment phase.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years of age or older.
2. Have a diagnosis of moderate-to-severe psoriasis for at least 6 months confirmed by a dermatologist, defined here as plaque-type psoriasis affecting a body surface area of >10% and a PASI of >10.
3. Agree to avoid prolonged sun exposure and avoid use of tanning booths or other ultraviolet light sources during the study.
4. Ability to understand and sign written informed consent.
5. Heterosexually active men and women of childbearing potential must use two methods of contraception during the study (20 weeks) and for 90 days after study completion. The two methods of birth control may be used simultaneously in the same subject or simultaneously in both partners. The two birth control methods can be (a) 2 barrier methods or (b) a barrier method plus a hormonal method to prevent pregnancy.

   Barrier methods include: condom (female or male), copper intrauterine device, sponge, or spermicide.

   Hormonal Methods include: any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent, including oral, subcutaneous, intrauterine, or intramuscular agents.
6. For pre-menopausal women, a negative pregnancy test, obtained within 1 week prior to first study drug dose and at study visits Week 0, Week 6, Week10, Week 14, and Week 20. If at any visit during the Treatment Phase (see Appendix A) a positive pregnancy test is returned, the subject will be discontinued from any further study drug.
7. Negative serology for human immunodeficiency virus 1 and 2 (HIV1/2), hepatitis B and hepatitis C.
8. The following screening laboratory blood tests must have the following values, or not clinically significant as determined by the PI and Medical Monitor: white blood cells (WBC) within normal limits (WNL); absolute neutrophil count > lower limit of normal; platelet count WNL; hemoglobin >10.0 g/dL; aspartate aminotransferase (AST) < 2.5 x the upper limit of normal.
9. Adequate renal function: creatinine clearance estimated by Cockcroft-Gault formula >60 ml/min

Exclusion Criteria:

1. Known history of hepatitis, HIV infection, interstitial lung disease.
2. Greater than moderate alcohol consumption on a regular basis (moderate consumption for females is 1 drink or 1 glass of wine a day; for males is 2 drinks or 2 glasses of wine a day) and unwilling, or unable, to control consumption during the study period.
3. Prior use of aminopterin (AMT).
4. Use of these biologic treatments in the time frames specified:

   * Within 9 months of first study drug dose: ustekinumab (Stelara).
   * Within 12 weeks of first study drug dose: any experimental therapy for psoriasis or rheumatoid arthritis.
   * Within 8 weeks of first study drug dose: infliximab (Remicade), adalimumab (Humira).
   * Within 4 weeks of first study drug dose: etanercept (Enbrel).
   * Other biologic therapies will have discontinuation periods determined by 5x their half-life.
5. Within 90 days prior to Day 0 and at any time while on study, the use of MTX.
6. Within 4 weeks prior to randomization and at any time while on study, use of phototherapy (e.g., ultraviolet B (UVB), narrow band UVB, Goeckerman regimen, Ingram regimen, PUVA), systemic medications (e.g. acitretin, mycophenolate mofetil, tacrolimus/FK506, cyclosporine A, azathioprine, 6-thioguanine, sulfasalazine, hydroxyurea, calcitriol, any systemic immunosuppressants), lithium, or any treatments that could affect psoriasis or sPGA evaluations. Subjects are eligible 4 weeks after the last dose of any of the aforementioned treatments was received.
7. Within 2 weeks prior to randomization and at any time while on study, use of any topical medications or treatments that could affect psoriasis evaluations (e.g., corticosteroids, anthralin, vitamin D3/calcitriol and analogues such calcipotriene and tacalcitol, synthetic retinoids such as tazarotene, coal tar, and keratolytics such as salicylic acid, lactic acid and urea including those contained in over-the-counter medicated shampoos). Subjects are eligible 2 weeks after the last dose of any of the aforementioned treatments was received.

   Note: Over-the-counter topical steroids will be permitted for use limited to the face, axilla, and/or genitalia, as needed. These topical medications should not be used within approximately 24 hours prior to study visits Day 0 and Day 98. Over-the-counter shampoos for the treatment of psoriasis of the scalp are also permitted.
8. Use of emollients on the morning of the first (Week 0) study visit.
9. Within 2 weeks prior to Study Day 0, or on Study Day 0, or at any time during the study, use of any of the following medications that may result in drug/drug interactions with AMT: trimethoprim with or without sulfamethoxazole; sulfonamides; sulfonylureas; pyrimethamine; tromethamine; salicylates; non-steroidal anti-inflammatory (NSAID) drugs including ibuprofen; dipyridamole; colchicine; probenecid; aminoglycosides; theophylline; phenytoin; and folinic acid (i.e., leucovorin).
10. Known concurrent malignancy except basal or squamous cell skin carcinoma, or cervical carcinoma in situ.
11. Concurrent participation in another clinical trial involving experimental treatment within 30 days of Study Day 0.
12. Current and uncontrolled infection, cardiovascular, renal, pulmonary, hepatic or GI conditions that will interfere with the conduct of the trial or pose a morbid risk.
13. Investigator's opinion that a concurrent disease or condition impairs the subject's ability to complete the trial: includes psychological, familial, sociological, geographical or medical conditions.
14. Breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Kahn, MD, Study Director — Syntrix Biosystems
Locations (3):
- United States (3):
  - Spectrum Dermatology, Scottsdale, Arizona
  - Dermatology Associates of Seattle, Seattle, Washington
  - Premier Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Menter A, Thrash B, Cherian C, Matherly LH, Wang L, Gangjee A, Morgan JR, Maeda DY, Schuler AD, Kahn SJ, Zebala JA. Intestinal transport of aminopterin enantiomers in dogs and humans with psoriasis is stereoselective: evidence for a mechanism involving the proton-coupled folate transporter. J Pharmacol Exp Ther. 2012 Sep;342(3):696-708. doi: 10.1124/jpet.112.195479. Epub 2012 May 31. PMID 22653877

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LD-Aminopterin Oral Capsule | Placebo Oral Capsule
Started | 11 | 8
Completed | 8 | 6
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LD-Aminopterin Oral Capsule | Placebo Oral Capsule | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (10.3) | 50.0 (13.1) | 50.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 10 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 10 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 7 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Subjects With >=75% Reduction in Baseline Psoriasis Area and Severity Index (PASI) (Efficacy)
Description: As follows:
  1. Area of Involvement. Determine a score, from 0 to 6, for each body section (head, trunk, upper limbs, lower limbs) based on the percent of psoriasis skin involvement: 0=0%, 1=<10%, 2=10% to <30%, 3=30% to <50%, 4=50% to <70%, 5=70% to <90%, 6=90% to 100%.
  2. Severity of Involvement. Determine a score, from 0 to 4, for each body section (head, trunk, upper limbs, lower limbs), for the psoriatic skin severity of each of erythema, thickness, and scaling: 0=none, 1=slight, 2=moderate, 3=severe, 4=very severe. For each body section the three severity scores are summed.
  3. For each body section the product of the Area and Severity is determined.
  4. For each body section the product of line 3 is multiplied by an Area Factor (head=0.1, trunk=0.3, upper limbs=0.2, lower limbs=0.4).
  5. A PASI score is determined by summing the 4 body section products (line 4). The highest possible score=72; the lowest possible score=0. The higher the scores, the worse the psoriasis.
Time Frame: 98 days.
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | LD-Aminopterin Oral Capsule | Placebo Oral Capsule
Number analyzed (Participants) | 11 | 8
Participants | 3 | 1
Statistical Analysis 1: Comparison: LD-Aminopterin Oral Capsule vs Placebo Oral Capsule; The efficacy of LD-AMT established using a step-down analysis approach with one-sided Fisher's exact tests. First, the analysis for subjects attaining PASI 75 will be performed, then, if that analysis shows a significant treatment effect, analysis for subjects attaining a sPGA success will be performed; Test type: Superiority; p = 0.43, Fisher Exact

2. Primary Outcome: Success (Score of 0 or 1) in Static Physician Global Assessment (sPGA) (Efficacy)
Description: As follows:
  1. Induration. A score, from 0 to 5, based on: 0=No plaque elevation; 1= Minimal plaque elevation=0.25 mm; 2=Mild plaque elevation=0.5 mm; 3=Moderate plaque elevation=0.75 mm; 4=Marked plaque elevation=1.0 mm; 5=Severe plaque elevation>1.25 mm.
  2. Erythema. A score, from 0 to 5, based on: 0=No erythema, hyperpigmentation may be present; 1=Faint erythema; 2=Light red coloration; 3=Moderate red coloration; 4=Bright red coloration; 5=Dusky to deep red coloration.
  3. Scaling. A score, from 0 to 5, based on: 0= No scaling; 1=Minimal; occasional fine scale on<5% of the lesion; 2=Mild; fine scale predominates; 3=Moderate; coarse scale predominates; 4=Marked; thick, non-tenacious scale predominates; 5=Severe; very thick, tenacious scale predominates.
  4. The sPGA: Induration, Erythema, and Scaling scores are rounded to the nearest whole number and averaged. 0=Cleared; 1=Minimal; 2=Mild; 3=Moderate; 4=Marked; 5=Severe. Higher score indicates worse psoriasis.
Time Frame: 98 days.
Measure: Count of Participants; unit: Participants
Arm/Group | LD-Aminopterin Oral Capsule | Placebo Oral Capsule
Number analyzed (Participants) | 11 | 8
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 98 days will on treatment and 42 days afterward (140 days total)
Arm/Group | LD-Aminopterin Oral Capsule | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/8
Other Adverse Events (participants affected / at risk) | 5/11 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LD-Aminopterin Oral Capsule (N=11) | Placebo Oral Capsule (N=8)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) — Possibly related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LD-Aminopterin Oral Capsule (N=11) | Placebo Oral Capsule (N=8)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall retain title to and the right to publish all documentation, records, raw data, specimens or other work product generated in connection with the performance of the Services. Such publications shall not be made by PI without the prior written consent of Sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT03431974/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (Detailed) (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT03431974/SAP_001.pdf